CLINICAL TRIAL: NCT02393157
Title: Chemoimmunotherapy With Obinutuzumab, Ifosfamide, Carboplatin and Etoposide (O-ICE) in Children, Adolescents and Young Adults With Recurrent Refractory CD20+ Mature B-NHL
Brief Title: Obinutuzumab and ICE Chemotherapy in Refractory/Recurrent CD20+ Mature NHL
Acronym: O-ICE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: Roswell Park Cancer Institute (Other)
Responsible Party: Principal Investigator, Mitchell Cairo, Vice Chair, New York Medical College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-11,392
Record Dates: First submitted 2015-03-08; First posted 2015-03-19 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Non-Hodgkin Lymphoma; Burkitt Lymphoma; Diffuse Large B-Cell Lymphoma; Primary Mediastinal B-cell Lymphoma; CD20+ Lymphoblastic Lymphoma; Follicular Lymphoma, Grade III
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — obinutuzumab; Ifosfamide; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Central Nervous System (CNS) Negative (Experimental): All patients will receive 4 doses of obinutuzumab on days -14, -10, -6 and -2. Patients without CNS involvement will receive one dose of Liposomal cytarabine for CNS prophylaxis on day -13. Dexamethasone will be given for 5 days with each Liposomal cytarabine dose starting one day prior to the Liposomal cytarabine. Dexamethasone 0.15 mg/kg/dose (max 4mg) IV BID will be given days -14 to -10. Following completion of the Prephase (or at the first sign of progressive disease), all patients will proceed to cycle 1 of O-ICE. O-ICE chemotherapy is given in 21-day (3-week) cycles. Three weekly doses of obinutuzumab will be given days -2 (during the prephase), +6 and +13. Patients will receive ICE chemotherapy (ifosfamide-carboplatin-etoposide) administered on Days 0-2 of Cycle 1.
  Interventions: Drug: Obinutuzumab; Drug: Liposomal ARA-C; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide
- CNS Positive (Experimental): All patients will receive 4 doses of obinutuzumab on days -14, -10, -6 and -2. Patients with positive CSF prior to enrollment will receive treatment with two doses of Liposomal cytarabine during the prephase portion of therapy. Liposomal cytarabine will be given intrathecally on days -13 and -5. Dexamethasone will be given for 5 days with each Liposomal cytarabine dose starting the day prior to the Liposomal cytarabine. Dexamethasone will be given days -14 to -10 and days -6 through -2. Following completion of the Prephase (or at the first sign of progressive disease), all patients will proceed to cycle 1 of O-ICE. O-ICE chemotherapy is given in 21-day (3-week) cycles. Three weekly doses of obinutuzumab will be given days -2 (during the prephase), +6 and +13. Patients will receive ICE chemotherapy (ifosfamide-carboplatin-etoposide) administered on Days 0-2 of Cycle 1.
  Interventions: Drug: Obinutuzumab; Drug: Liposomal ARA-C; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Obinutuzumab — Drug will be given alone in a pre-phase and in combination with ICE chemotherapy.
  Other Names: Gazyva
Drug: Liposomal ARA-C — Will be given intrathecally for both prophylaxis and treatment of CNS disease.
  Other Names: Depocyte
Drug: Ifosfamide — Ifosfamide 3000 mg/m2/day as a 2 hour IV infusion daily x 3 days (Days 0,1,2) of Cycle 1 and 2.
  Other Names: Ifex
Drug: Carboplatin — Carboplatin: 635 mg/m2 as 1 hour IV infusion on Day 0 only of Cycle 1 and 2.
  Other Names: Paraplatin
Drug: Etoposide — Etoposide: 100 mg/m2/day as 1 hour IV infusion daily x 3 days (Days 0,1,2).
  Other Names: VP-16

SUMMARY:
The purpose of this study is to determine the safety of administering obinutuzumab as a single agent alone and in combination with ifosfamide, carboplatin, and etoposide (ICE) chemotherapy and determine the response rate of this treatment for children, adolescents and young adults (CAYA) with relapsed CD20 positive B-cell Non-Hodgkin Lymphoma (B-NHL).

ELIGIBILITY:
Inclusion Criteria:

* Patients in first relapse or primary induction failure CD20 positive B-cell leukemia/lymphoma including:

  * Diffuse Large B-Cell Lymphoma
  * Burkitt Lymphoma
  * High Grade B-cell Lymphoma: Not Otherwise Specified (NOS)
  * Primary mediastinal B-cell lymphoma (PMBL)
  * CD20+ B-lymphoblastic lymphoma
  * Follicular lymphoma, Grade III
  * Karnofsky ≥ 60% for patients > 16 years of age and
  * Lansky ≥ 60 for patients ≤ 16 years of age.
  * Myelosuppressive chemotherapy: Must not have received within 2 weeks of entry onto this study.
  * Patients may not have received prior therapy with obinutuzumab (GA101)
  * Radiation Therapy (XRT): Date of receiving prior XRT must be > 2 weeks for local palliative XRT (small port); > 6 months must have elapsed if prior craniospinal XRT or if > 50% radiation of pelvis; > 6 weeks must have elapsed if other substantial bone marrow radiation.
  * Steroids: Patients may have received prior steroid treatment, but not started greater than 7 days prior to initiation of protocol therapy.
  * Adequate organ function.

Exclusion Criteria:

* Patients with newly diagnosed, previously untreated B-NHL.
* Known congenital or acquired immune deficiency.
* Prior solid organ transplantation.
* Prior allogeneic stem cell transplant within 60 days or active acute Graft-vs-Host-Disease (GVHD) grade 3 or higher.
* History of grade 4 anaphylactic reactions to humanized or murine monoclonal antibodies
* Uncontrolled hepatitis B and/or C infection

Ages: 3 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-08-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by adverse reactions and events | 1 month
  Patients will be monitored for adverse reactions and events of drug when given alone and in combination with ICE chemotherapy.
Response rate assessed following each treatment cycle for regression of tumor | 3 months
  Patients will be assessed following each treatment cycle for regression of tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD, Study Chair — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States